CLINICAL TRIAL: NCT00257881
Title: Phase 1 Dose-Escalation Study of Intravenous CMD-193 in Subjects With Advanced Malignant Solid Tumors
Brief Title: Study Evaluating Intravenous CMD-193 in Subjects With Advanced Malignant Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3152K1-101
Record Dates: First submitted 2005-11-22; First posted 2005-11-23 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Neoplasms
Keywords: Tumor
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Drug: CMD-193

SUMMARY:
The primary purpose of this study is to evaluate the safety, tolerability, and maximum tolerated dose (MTD) of CMD-193 administered intravenously (IV) to subjects with advanced malignant tumors. The secondary purpose is to obtain preliminary information on the pharmacokinetics and antitumor activity of IV CMD-193.

ELIGIBILITY:
Inclusion Criteria:

* Malignant solid tumor progressed, or no standard treatment available
* Tumor expression of Lewis Y antigen

Exclusion Criteria:

* Cancer therapy within 28 days before enrollment
* Pregnant or breastfeeding women
* Unstable or serious concurrent medical conditions

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46
Dates: Start 2005-11; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity, Adverse Event

SECONDARY OUTCOMES:
Pharmacokinetics parameters, Tumor assessment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (2):
- Japan (2):
  - Tokyo, Chuo-ku
  - Nagaizumi-cho, Sunto-gun, Shizuoka